CLINICAL TRIAL: NCT00152594
Title: Phase III Study of Safety, Tolerance, Efficacy, Pharmacokinetics, and Costs of Therapy With Voriconazole or Placebo in the Prophylaxis of Lung Infiltrates in Patients Undergoing Induction Chemotherapy for Acute Myelogenous Leukemia
Brief Title: Voriconazole or Placebo in the Prophylaxis of Lung Infiltrates in Patients Undergoing Induction Chemotherapy for Acute Myelogenous Leukemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cologne (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NRA 150 0009
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2006-11-14 (Estimated); Status verified 2006-11

CONDITIONS: Leukemia, Myelocytic, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Voriconazole

INTERVENTIONS:
Drug: voriconazole

SUMMARY:
The purpose of the study is to determine whether voriconazole is as effective as antifungal prophylaxis in patients undergoing chemotherapy for acute myelogenous leukemia (AML).

Hypothesis: Voriconazole is superior to placebo in the prophylaxis of lung infiltrates until day 21 after the start of induction chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed or relapsed, de novo or secondary AML
2. First induction chemotherapy cycle
3. Expected neutropenic phase of a minimum duration of 10 days
4. Age >= 18 years
5. Legally signed consent form

Exclusion Criteria:

1. Known proven, probable or possible invasive fungal infection at randomization or in patient history
2. Computed tomography (CT) with any signs of a fungal infection according to the European Organisation for the Research and Treatment of Cancer (EORTC)/Mycosis Study Group (MSG) criteria, i.e. with any infiltrate (Ascioglu, et al 2002)
3. Any current fever unless explained by non-infectious causes
4. Antibacterial prophylaxis other than TMP/SMX
5. Liver function test [LFT] (AST/ALT/bilirubin) more than 3x the upper normal limit
6. Subjects who are receiving and cannot discontinue one of the following drugs at least 24 hours prior to randomization:

   * Drugs with a known possibility of QTc prolongation (e.g. terfenadine, astemizole, cisapride, pimozide, quinidine);
   * Drugs whose plasma levels may be increased by voriconazole therapy (e.g. sulfonylureas, ergot alkaloids, sirolimus, vinca alkaloids).
7. Subjects who have received the following drugs within 14 days prior to randomization: potent inducers of hepatic enzymes that will reduce voriconazole levels (e.g. rifampicin, carbamazepine and barbiturates)
8. Concomitant therapy with absorbable antifungals
9. Patient has a diagnosis of acute hepatitis or cirrhosis due to any cause
10. Known hypersensitivity or other contraindication to voriconazole
11. Patient is unwilling or unable to comply with the protocol.
12. Diseases or disabilities preventing the patient from participating in the trial
13. Females of childbearing potential without negative serum pregnancy test at baseline or within 72 hours prior to start of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2004-10; Study Completion 2006-01

PRIMARY OUTCOMES:
To determine the incidence of lung infiltrates until day 21 among patients undergoing the first induction chemotherapy for acute myelogenous leukemia who are randomized to prophylactic voriconazole or placebo

SECONDARY OUTCOMES:
To determine and compare between study arms the: incidence of fever and other signs of infection
incidence and type of documented bacteremia
rate of patients with systemic open-label antifungal therapy
time to initiation of systemic open-label antifungal therapy
duration of absolute neutrophil count < 500/µl
rate and type of proven, probable and possible breakthrough invasive fungal infections
rate of patients with fever of unknown origin
incidence and severity of adverse events
trough voriconazole plasma level after day 8 of study treatment
direct costs of systemic antibiotics, antifungals and antivirals and diagnostic imaging
overall costs in terms of the diagnosis related groups applied to the study patients

CONTACTS AND LOCATIONS:
Overall Officials: Oliver A. Cornely, MD, Principal Investigator — Klinikum der Universität Köln
Locations (3):
- Germany (3):
  - Klinikum der Universität Köln, Cologne
  - Johann Wolfgang Goethe-Universität Frankfurt am Main, Frankfurt am Main
  - Universitätsklinikum Mannheim, Universität Heidelberg, Heidelberg